CLINICAL TRIAL: NCT02485548
Title: A Multicenter Phase Ⅲ Trial of Cisplatin Plus Raltitrexed or 5-fluorouracil in Concurrence With Intensity-modulated Radiotherapy (IMRT) for the Treatment of Locoregionally Advanced Head and Neck Squamous Cell Cancer
Brief Title: Cisplatin Plus Raltitrexed or 5-fluorouracil Concurrent With Radiotherapy for Head and Neck Squamous Cell Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Collaborators: Affiliated Hospital of Jiangnan University (Other); Changzhou Cancer Hospital of Soochow University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Northern Jiangsu People's Hospital (Other); The Second Hospital of Nanjing Medical University (Other); Nanjing BenQ Hospital (Unknown)
Responsible Party: Principal Investigator, Dr. Xia He, Director of Radiation Oncology, Jiangsu Cancer Institute & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014NL-035
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Head and Neck Squamous Cell Cancer
MeSH Terms: interventions — raltitrexed; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltitrexed plus cisplatin (Experimental): Raltitrexed plus cisplatin and IMRT
  Interventions: Drug: Raltitrexed; Drug: Cisplatin; Radiation: IMRT
- 5-fluorouracil plus cisplatin (Active Comparator): 5-fluorouracil plus cisplatin and IMRT
  Interventions: Drug: 5-fluorouracil; Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: Raltitrexed — Patients will receive IMRT and concurrent raltitrexed and cisplatin
  Arms: Raltitrexed plus cisplatin
Drug: 5-fluorouracil — Patients will receive IMRT and concurrent 5-Fu and cisplatin
  Arms: 5-fluorouracil plus cisplatin
Drug: Cisplatin — All patients will receive concurrent cisplatin.
Radiation: IMRT — All patients will receive IMRT

SUMMARY:
This study is a multicenter phase Ⅲ trial. The objective is to compare the efficacy and toxicity of cisplatin plus raltitrexed or 5-fluorouracil in concurrence with IMRT for patients with locoregionally advanced head and neck squamous cell cancer.

DETAILED DESCRIPTION:
The objective is to compare the efficacy and toxicity of cisplatin plus raltitrexed or 5-fluorouracil in concurrence with IMRT for patients with locoregionally advanced head and neck squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed untreated head and neck squamous cell cancer patients
* 18-70 years
* Clinical stage: T3-4N0-3M0 or T1-4N1-3M0
* Hematologic function: WBC ≥ 4.0×109/L, PLT ≥ 80×109/L, Hb ≥ 10mg/dL
* Renal function: Cr ≤ 1.25×UNL
* Hepatic function: BIL ≤ 1.5×UNL, ALT/AST ≤ 2.5×UNL
* ECOG ≤ 1
* Woman and man of childbearing age must adopt contraception
* With written consent

Exclusion Criteria:

* Malignant history
* Pregnant or lactating women
* With other severe diseases (blood, liver ,kidney or heart diseases)
* Subjects not suitable for chemo-radiotherapy
* Without written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 36 months

SECONDARY OUTCOMES:
Overall Survival (OS) | 36 months
Locoregional and distant control rate | 36 months
Percentage of participants experiencing grade 3-5 adverse events(AEs) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Xia He, M.D., Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China